CLINICAL TRIAL: NCT02749747
Title: Sulpiride Versus Placebo for Reducting Hot Flushes During Climacteric: a Double-blind Randomized Clinical Trial
Brief Title: Sulpiride Versus Placebo for Reducting Hot Flushes During Climacteric
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0038
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2018-01

CONDITIONS: Menopausal Syndrome; Hot Flashes
Keywords: Menopause; nonhormonal treatment; sulpiride
MeSH Terms: conditions — Hot Flashes | interventions — Sulpiride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sulpiride use (Active Comparator): 50mg sulpiride once a day use for 60 days
  Interventions: Drug: Sulpiride use
- Placebo (Placebo Comparator): 50mg placebo once a day use for 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulpiride use — 50mg sulpiride once a day use for 60 days
  Other Names: Sulpirida
  Arms: Sulpiride use
Drug: Placebo — 50mg placebo once a day use for 60 days
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
* Introduction: Estrogen hormonal therapy associated or not with progestagen is the standard therapy for the treatment of hot flushes. However some women are not candidates for hormone replacement therapy for medical reasons or for choice.
* Main goal: Reducing the number of hot flushes per week
* Materials and Methods: A double-blind sulpiride versus placebo that includes selected randomized patients which show symptoms of menopause. The study will be conducted at HC Porto Alegre (Brazil) for 8 weeks of intervention. The expected result is a significant reduction in the number of hot flushes/day evaluated by daily questionnaires

DETAILED DESCRIPTION:
It will be held 4 visits. The V0 (first one) to implement the consent form, review the inclusion and exclusion criteria and laboratory exams and deliver the diary book of hot flushes. The V1 (second visit) randomization and provide medication for the first 30 days. The V2 (third visit) to make the record diary of hot flushes already filled, to deliver new specifications and to provide medication for the last 30 days. The V3 (fourth visit) to evaluate the record diary of hot flushes already completed and to make a final evaluation of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women in postmenopausal women with at least five moderate to intense hot flushes per day

Exclusion Criteria:

* Use of hormone replacement therapy or psychiatric drugs for at least 3 months
* Hypersensitivity to sulpiride
* Current or history of prolactin dependent tumor
* Treating breast cancer or treated
* Diagnosed or suspected pheochromocytoma
* Current use of levodopa
* Abnormal heart rhythm (QT prolongation, bradycardia low 55 beats per minute)
* Hypokalemia and other serious electrolyte disturbances
* Current or treated stroke
* Pregnancy or breastfeeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number and severity records of hot flushes | From baseline to eight weeks
  Daily diary of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Maria Celeste Osorio Wender, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pedro AO, Pinto Neto AM, Paiva LH, Osis MJ, Hardy E. [Age at natural menopause among Brazilian women: results from a population-based survey]. Cad Saude Publica. 2003 Jan-Feb;19(1):17-25. doi: 10.1590/s0102-311x2003000100003. Epub 2003 Apr 1. Portuguese. PMID 12700780
- [Background] Vilodre LC, Moretto M, Kohek MB, Spritzer PM. [Premature ovarian failure: present aspects]. Arq Bras Endocrinol Metabol. 2007 Aug;51(6):920-9. doi: 10.1590/s0004-27302007000600005. Portuguese. PMID 17934658
- [Background] De Lorenzi DR, Baracat EC, Saciloto B, Padilha I Jr. [Factors related to quality of life in post-menopause]. Rev Assoc Med Bras (1992). 2006 Sep-Oct;52(5):312-7. doi: 10.1590/s0104-42302006000500017. Portuguese. PMID 17160304
- [Background] Wender, M.C. et al. Consenso Brasileiro de Terapêutica Hormonal da Menopausa. SOBRAC - Leitura Médica. 2014.
- [Background] Oderich, C. L., Wender, M.C. Climatério. Revista Brasileira de Medicina. 69, 2012.
- [Result] Sussman M, Trocio J, Best C, Mirkin S, Bushmakin AG, Yood R, Friedman M, Menzin J, Louie M. Prevalence of menopausal symptoms among mid-life women: findings from electronic medical records. BMC Womens Health. 2015 Aug 13;15:58. doi: 10.1186/s12905-015-0217-y. PMID 26271251
- [Result] Boardman HM, Hartley L, Eisinga A, Main C, Roque i Figuls M, Bonfill Cosp X, Gabriel Sanchez R, Knight B. Hormone therapy for preventing cardiovascular disease in post-menopausal women. Cochrane Database Syst Rev. 2015 Mar 10;2015(3):CD002229. doi: 10.1002/14651858.CD002229.pub4. PMID 25754617
- [Result] Loprinzi CL, Stearns V, Barton D. Centrally active nonhormonal hot flash therapies. Am J Med. 2005 Dec 19;118 Suppl 12B:118-23. doi: 10.1016/j.amjmed.2005.09.045. PMID 16414336
- [Result] Carroll DG, Lisenby KM, Carter TL. Critical appraisal of paroxetine for the treatment of vasomotor symptoms. Int J Womens Health. 2015 Jun 18;7:615-24. doi: 10.2147/IJWH.S50804. eCollection 2015. PMID 26124682
- [Result] Umland EM, Falconieri L. Treatment options for vasomotor symptoms in menopause: focus on desvenlafaxine. Int J Womens Health. 2012;4:305-19. doi: 10.2147/IJWH.S24614. Epub 2012 Jul 5. PMID 22870045
- [Result] Pachman DR, Jones JM, Loprinzi CL. Management of menopause-associated vasomotor symptoms: Current treatment options, challenges and future directions. Int J Womens Health. 2010 Aug 9;2:123-35. doi: 10.2147/ijwh.s7721. PMID 21072305
- [Result] Bruscky SB, Caldeira MV, Bueno JR. [Clinical trial with sulpiride]. Arq Neuropsiquiatr. 1974 Sep;32(3):234-9. doi: 10.1590/s0004-282x1974000300010. No abstract available. Portuguese. PMID 4408939
- [Result] Simon JA, Chandler J, Gottesdiener K, Lazarus N, He W, Rosenberg E, Wagner JA, Denker AE. Diary of hot flashes reported upon occurrence: results of a randomized double-blind study of raloxifene, placebo, and paroxetine. Menopause. 2014 Sep;21(9):938-44. doi: 10.1097/GME.0000000000000218. PMID 24569618